CLINICAL TRIAL: NCT01341301
Title: A Two Step Approach to Allogeneic Hematopoietic Stem Cell Transplantation for High-Risk Hematologic Malignancies Using One Human Leukocyte Antigen Partially-Matched Related Donor
Brief Title: Donor Stem Cell Transplant in Treating Patients With High-Risk Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10D.06; 2009-41 (Other: CCRRC); JT 1521 (Other: JeffTrial Number)
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hematologic Malignancy
Keywords: allogeneic stem cell transplant; TJU 2 Step; HSCT; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Whole-Body Irradiation; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic HSCT (Experimental): CONDITIONING: Patients undergo Total Body Irradiation (TBI) twice daily (BID) on days -10 to -7. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients receive DLI on day -6 and undergo cluster of differentiation 34 (CD34+) selected allogeneic HSCT on day 0
  GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO on days -1 with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID or PO on days -1 to 28.
  Interventions: Radiation: Total Body Irradiation; Biological: Donor Lymphocyte Infusion (DLI); Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Procedure: Allogeneic hematopoietic stem cell transplantation; Other: Laboratory biomarker analysis

INTERVENTIONS:
Radiation: Total Body Irradiation — Undergo TBI
  Other Names: TBI
Biological: Donor Lymphocyte Infusion (DLI) — Undergo DLI
  Other Names: DLI
Drug: Cyclophosphamide — Given IV
  Other Names: Cytoxan; Endoxan; Endoxana; Enduxan
Drug: Tacrolimus — Given IV or PO
  Other Names: Advagraf; Prograf; Protopic
Drug: Mycophenolate mofetil — Given IV or PO
  Other Names: Cellcept
Procedure: Allogeneic hematopoietic stem cell transplantation — Undergo allogeneic HSCT
Other: Laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this research study is to examine the survival of patients undergoing partially matched hematopoietic stem cell transplant (HSCT) on a new type of treatment approach, which has been developed specifically for patients who have evidence of their disease at the time of transplant. In this research study, a way of strengthening the response of the donor cells against the disease has been developed. Patients will undergo one additional day between the two steps of the transplant which may allow their donor's cells to fight the disease more effectively.

DETAILED DESCRIPTION:
This is a phase II study in which patients receive a haploidentical HSCT from a single donor. The period between the donor lymphocyte infusion (DLI) and tolerizing doses of CY has been extended to allow for an increased period of allogeneic response against tumor targets. The outcomes of patients undergoing this extra time period will be compared to historical data to assess efficacy.

Primary Objective:

1) To assess 1 year relapse free survival in patients undergoing hematopoietic stem cell transplant (HSCT) using the Thomas Jefferson University (TJU) 2 step approach with an extra day inserted between the DLI and administration of cyclophosphamide (CY).

Secondary Objectives:

1. To assess the consistency and pace of engraftment.
2. To assess the pace of T cell and B cell immune recovery.
3. To assess regimen related toxicity, (GVHD) graft-versus-host disease incidence and severity, and overall survival in patients undergoing treatment on this protocol. .
4. To assess the tolerance of the period of fever, diarrhea, and rash in each arm in an effort to determine whether a longer interval prior to cytoxan changes this side effect qualitatively compared to prior patient groups or concurrent patient groups. N.B. Patients with hematologic malignancies in remission will continue to be transplanted without modification to the original 2-step approach and will serve as a concurrent comparison group.
5. To collect leukemia samples prior to transplant and after relapse whenever possible. To assess the overall degree of HLA-class I and class II expression on these paired samples. To test for loss of one or both HLA haplotypes in the relapsed tumor specimens.
6. To determine the number of cluster of differentiation 4 (CD4+) cluster of differentiation 25 (CD25+) FOXP3+ regulatory cells post HSCT and to assess whether this is correlated with the development of GVHD after transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a hematologic malignancy with residual disease after treatment with 1 or more chemotherapy regimens in whom achievement of remission with additional chemoradiotherapy is felt to be unlikely or who is in 3rd or greater complete remission (CR).

   Patients with marrow based diseases in which the marrow biopsy does not meet criteria for active disease (ie <5% blasts in acute leukemia) but who does not have full count recovery will be eligible for treatment on this high risk trial.
2. Patients must have at least one related donor who is HLA mismatched in the GVHD direction at two or more HLA loci.
3. Patients must adequate organ function:

   1. Left ventricular ejection fraction (LVEF) of >50 %
   2. Diffusion capacity of the lung for carbon monoxide (DLCO) (adjusted for hemoglobin) >50 % of predicted
   3. Adequate liver function as defined by a serum bilirubin <1.8, Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2.5 times upper limit of normal
   4. Creatinine clearance of > 60 ml/min
4. Karnofsky Performance Status of > 80% on the modified KPS tool
5. Patients must be willing to use contraception if they have childbearing potential.
6. Able to give informed consent

Exclusion Criteria:

1. Modified Karnofsky performance status (KPS) of <80%
2. > 5 Comorbidity Points on the hematopoietic cell transplantation comorbidity index (HCT-CI) Index
3. Untreated class I or II antibodies against donor HLA antigens
4. HIV positive
5. Active involvement of the central nervous system with malignancy
6. Psychiatric disorder that would preclude patients from signing an informed consent
7. Pregnancy, or unwillingness to use contraception if they have child bearing potential
8. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder
9. Alemtuzumab treatment within 8 weeks of HSCT admission.
10. Anti-thymocyte globulin (ATG) level of > 2 ugm/ml
11. Patients with active inflammatory processes including Tmax >101 or active tissue inflammation are excluded
12. Inability to tolerate cyclophosphamide or undergo total body irradiation at the doses specified in the treatment plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05; Primary Completion 2013-11-04 (Actual); Study Completion 2014-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Principal Investigator — Thomas Jefferson University; Dolores Grosso, DNP, CRNP, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Allogeneic HSCT: CONDITIONING: Patients undergo total body irradiation (TBI) twice daily (BID) on days -10 to -7. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients receive Donor Lymphocyte Infusion (DLI) on day -6 and undergo cluster of differentiation (CD34+) selected allogeneic HSCT on day 0
  Graft-versus-host disease (GVHD) PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO on days -1 with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID or PO on days -1 to 28.
  Total Body Irradiation: Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Tacrolimus: Given IV or PO
  Mycophenolate mofetil: Given IV or PO
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  Laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Allogeneic HSCT
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Allogeneic HSCT: CONDITIONING: Patients undergo TBI BID on days -10 to -7. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients receive DLI on day -6 and undergo CD34+ selected allogeneic HSCT on day 0
  GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO on days -1 with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID or PO on days -1 to 28.
  Total Body Irradiation: Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Tacrolimus: Given IV or PO
  Mycophenolate mofetil: Given IV or PO
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  Laboratory biomarker analysis: Correlative studies
Arm/Group | Allogeneic HSCT
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience One Year Relapse Free Survival After Undergoing Hematopoietic Stem Cell Transplant (HSCT)
Description: To assess relapse free survival in participants undergoing Hematopoietic Stem Cell Transplant (HSCT) using the Thomas Jefferson University 2 step approach with an extra day inserted between the donor lymphocyte infusion (DLI) and administration of cyclophosphamide.
Time Frame: 1 year after undergoing hematopoietic stem cell transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic HSCT
Number analyzed (Participants) | 25
Participants | 5

2. Secondary Outcome: Pace of T-cell and B-cell Immune Recovery
Description: Reported descriptively
Time Frame: Assessed up to 1 year
Population: Data were not collected
Arm/Group | Allogeneic HSCT
Number analyzed (Participants) | 0

3. Secondary Outcome: Regimen Related Toxicities Graded According to the National Cancer Institute (NCI) Common Toxicity Criteria, Version 3.0
Description: Reported descriptively
Time Frame: Assessed up to 1 year
Population: Data were not collected
Groups:
- Allogeneic HSCT: CONDITIONING: Patients undergo Total Body Irradiation (TBI) twice daily (BID) on days -10 to -7. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients receive DLI on day -6 and undergo cluster of differentiation 34 (CD34+) selected allogeneic HSCT on day 0
  GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO on days -1 with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID or PO on days -1 to 28.
  Total Body Irradiation: Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Tacrolimus: Given IV or PO
  Mycophenolate mofetil: Given IV or PO
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  Laboratory biomarker analysis: Correlative studies
Arm/Group | Allogeneic HSCT
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence and Severity of GVHD, Graded According to Standard Criteria
Description: Reported descriptively
Time Frame: Assessed up to 1 year
Population: Data were not collected
Groups:
- Allogeneic HSCT: CONDITIONING: Patients undergo total body irradiation (TBI) twice daily (BID) on days -10 to -7. Patients also receive cyclophosphamide IV over 2 hours on days -3 and -2.
  TRANSPLANTATION: Patients receive DLI on day -6 and undergo cluster of differentiation (CD34+) selected allogeneic HSCT on day 0
  Graft-versus-host disease (GVHD) PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV or PO on days -1 with taper beginning on day 42. Patients also receive mycophenolate mofetil IV BID or PO on days -1 to 28.
  Total Body Irradiation: Undergo TBI
  Donor Lymphocyte Infusion (DLI): Undergo DLI
  Cyclophosphamide: Given IV
  Tacrolimus: Given IV or PO
  Mycophenolate mofetil: Given IV or PO
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic HSCT
  Laboratory biomarker analysis: Correlative studies
Arm/Group | Allogeneic HSCT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Allogeneic HSCT
Serious Adverse Events (participants affected / at risk) | 25/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HSCT (N=25)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 2 (2)
Agitation (General disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
CMV colitis (Gastrointestinal disorders) | 1 (1)
CMV reactivation (Gastrointestinal disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Elevated liver enzymes (Renal and urinary disorders) | 1 (1)
Fevers (General disorders) | 2 (3)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Hypoxia (Blood and lymphatic system disorders) | 4 (6)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Reintubation (General disorders) | 1 (1)
Respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Syncope (Blood and lymphatic system disorders) | 1 (1)
Volume overload (Ear and labyrinth disorders) | 1 (1)
Weight gain (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic HSCT (N=25)
Abdominal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2)
Abdominal pain (Musculoskeletal and connective tissue disorders) | 8 (10)
Abnormal LFTs (Renal and urinary disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Agitation (Musculoskeletal and connective tissue disorders) | 5 (5)
Ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 8 (9)
Aphasia (Nervous system disorders) | 1 (1)
Arm pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arm swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bacteremia (Blood and lymphatic system disorders) | 3 (4)
Benign prostatic hyperplasia (Renal and urinary disorders) | 1 (1)
BK viremia (Infections and infestations) | 2 (2)
Black eye (Eye disorders) | 1 (1)
Blister (General disorders) | 1 (1)
Blood-tinged sputum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blurry vision (Eye disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Calf pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Change in vision (Eye disorders) | 1 (1)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 5 (5)
Chills/rigors (General disorders) | 10 (12)
Clostridium difficile (Gastrointestinal disorders) | 1 (1)
CMV reactivation (General disorders) | 5 (5)
CMV viremia (Infections and infestations) | 1 (1)
Confusion (General disorders) | 5 (5)
Congestion (General disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7)
Cough (General disorders) | 8 (9)
Crackles (General disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5)
Decreased urine output (Renal and urinary disorders) | 2 (2)
Deep vein thrombosis (Cardiac disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Diaphoresis (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (21)
Difficulty breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Difficulty hearing (Ear and labyrinth disorders) | 1 (1)
Dizziness (General disorders) | 3 (3)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry mouth (General disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dysarthria (Cardiac disorders) | 1 (1)
Dysgeusia (General disorders) | 1 (1)
Dysphagia (General disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dysuria (Renal and urinary disorders) | 4 (4)
Edema (General disorders) | 12 (16)
Electrolyte imbalance (General disorders) | 6 (8)
Elevated alkaline phosphatase (General disorders) | 1 (1)
Elevated liver enzymes (Renal and urinary disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 2 (2)
Epistaxis (General disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2)
Eye dryness (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 9 (10)
Feet/ankle swelling (General disorders) | 2 (2)
Fevers (General disorders) | 17 (30)
Flank pain (General disorders) | 2 (2)
Gas pain (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
General pain (General disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 2 (2)
Hand/foot tightness (General disorders) | 1 (1)
Headache (General disorders) | 12 (17)
Hematoma (Blood and lymphatic system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (5)
Hemochromatosis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hernia (Gastrointestinal disorders) | 1 (1)
HHV6 viremia (Infections and infestations) | 3 (3)
Hiccups (General disorders) | 2 (2)
Hip pain (General disorders) | 2 (2)
Hives (General disorders) | 4 (4)
Hoarseness (General disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 8 (8)
Hypercholesterolemia (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Hives (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperglycemia (General disorders) | 1 (1)
Hyperkalemia (General disorders) | 1 (1)
Hypernatremia (Blood and lymphatic system disorders) | 2 (2)
Hypertension (General disorders) | 10 (12)
Hypervolemia (General disorders) | 5 (5)
Hypokalemia (General disorders) | 2 (3)
Hyponatremia (General disorders) | 2 (2)
Hypotension (General disorders) | 12 (14)
Hypoxia (General disorders) | 6 (6)
Increased creatinine (Blood and lymphatic system disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 2 (2)
Infection, other (Infections and infestations) | 2 (2)
Insomnia (General disorders) | 8 (8)
Intolerance to cold (General disorders) | 1 (1)
Itchiness (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (General disorders) | 1 (1)
Joint pain (General disorders) | 1 (1)
Leg tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Lethargy (General disorders) | 5 (5)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lip swelling (Skin and subcutaneous tissue disorders) | 2 (2)
Lung effusion (General disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Mental status change (Nervous system disorders) | 2 (2)
Metabolism disorder, other (Metabolism and nutrition disorders) | 3 (3)
Mucositis (General disorders) | 13 (13)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 20 (21)
Neck discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (General disorders) | 1 (1)
Neck swelling (General disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 3 (3)
Nocturia (General disorders) | 2 (2)
Non-ST segment elevation myocardial infarction (Cardiac disorders) | 1 (1)
Odynophagia (General disorders) | 2 (2)
Oral discomfort (General disorders) | 3 (3)
Oral pain (General disorders) | 2 (2)
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Parasthesia (General disorders) | 3 (3)
Parotid glad pain (General disorders) | 1 (1)
Pelvic pain (General disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pericatheter DVT (Vascular disorders) | 1 (1)
Peripheral edema (General disorders) | 1 (1)
Peri-rectal discomfort (General disorders) | 1 (1)
Petechia (Vascular disorders) | 1 (2)
Phlebitis (Vascular disorders) | 1 (1)
Pleural effusion (Vascular disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Polyneuromyopathy (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 15 (22)
Red eyes (Eye disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Restless leg (Nervous system disorders) | 1 (1)
Rhinorrhea (General disorders) | 1 (1)
Seizures (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sialadenitis (General disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
SIRS (General disorders) | 1 (1)
Skin pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin wound (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (General disorders) | 1 (1)
Sore on tip of penis (General disorders) | 1 (1)
Sore throat (General disorders) | 7 (7)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Supraventricular tachycardia (General disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 14 (17)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Tearing of eyes (Eye disorders) | 1 (1)
Temporal wasting (General disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrombus (Blood and lymphatic system disorders) | 1 (1)
Thrush (General disorders) | 1 (1)
Tongue pain (General disorders) | 2 (2)
Tracheal pain (General disorders) | 1 (1)
Transfusion reaction event (General disorders) | 1 (1)
Tremors (Nervous system disorders) | 3 (3)
Upper respiratory tract infection symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Urinary retention (Renal and urinary disorders) | 4 (4)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Ventricular trigeminy (Cardiac disorders) | 1 (1)
Vivid dreams (General disorders) | 1 (1)
Volume overload (General disorders) | 4 (4)
Vomiting (General disorders) | 7 (7)
Weakness (Nervous system disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes